CLINICAL TRIAL: NCT03883776
Title: Al18F-NOTA-octreotide PET Imaging of the Somatostatin Receptor in Neuroendocrine Tumors: a First-in-human PET/CT Study
Brief Title: Al18F-NOTA-octreotide PET Imaging of the Somatostatin Receptor in Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S61727
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Tumors
Keywords: PET/CT; Somatostatin receptor imaging; Al18F-NOTA-octreotide
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Al18F-NOTA-octreotide; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers and NET patients (Experimental): In the first part of the study, 6 healthy volunteers will receive a single intravenous single injection of Al18F-NOTA-octreotide, followed by whole-body PET/CT scans at various time points for an initial safety assessment and dosimetry study.
  In the second part of the study, a single dose of Al18F-NOTA-octreotide will be intravenously injected in 6 patients with neuroendocrine tumors. Patients will first undergo a dynamic PET scan, followed by whole-body PET/CT scans at various time points for a pharmacokinetics study and initial efficacy assessment.
  Interventions: Drug: Al18F-NOTA-octreotide; Device: PET/CT; Other: Venous blood samples

INTERVENTIONS:
Drug: Al18F-NOTA-octreotide — One intravenous injection of 4 MBq/kg
  Other Names: 18F-AlF-NOTA-octreotide; 18F-IMP-466
Device: PET/CT — Part 1: Healthy volunteers will undergo consecutive whole-body PET scans, including one low-dose CT, for the first 90 minutes. At 150 ± 15 min and 300 ± 30 min post injection two additional static whole-body PET/CT scans will be acquired.
  Part 2: Neuroendocrine tumor patients will undergo a dynamic PET scan for the first 45 minutes, followed by 3 static whole-body PET/CTs at 60 ± 10 min, 120 ± 30 min and 180 ± 30 min post injection.
Other: Venous blood samples — Blood samples will be obtained for laboratory safety evaluation for initial screening and safety evaluation after injection. Furthermore, venous blood samples will be obtained for metabolite analysis and activity measurements (only for patients) at various time points post injection (5 ± 2 min, 10 ± 5 min, 20 ± 10 min, 40 ± 20 min, 60 ± 30 min, 120 ± 60 min).

SUMMARY:
The aim of this study is to evaluate the potential of Al18F-1,4,7-triazacyclononane-1,4,7-triacetate-octreotide (Al18F-NOTA-octreotide) as a positron emission tomography (PET) somatostatin receptor imaging agent in patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
In the first part of the study, six healthy volunteers will undergo several sequential whole-body PET/CT scans starting from the moment of tracer injection up to six hours post injection for an initial safety assessment and dosimetry study of Al18F-NOTA-octreotide in humans.

In the second part of the study, six neuroendocrine tumor patients, with at least five positive lesions on routine clinical 68Ga-DOTA-peptide PET, will undergo a dynamic PET scan for the first 45 minutes, followed by three single static whole-body PET/CTs up to three hours post injection for an initial efficacy assessment (evaluation of the lesion detection rate) and pharmacokinetics study of Al18F-NOTA-octreotide in humans. Furthermore a first comparison with 68Ga-DOTA peptide PET will be performed.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Healthy volunteers:

* Age between 18 and 65 years
* Signed Informed Consent
* Subject is judged to be in good health by the investigator on the basis of medical history, physical examination including vital signs and clinical laboratory tests
* Female subjects should be post-menopausal or surgically sterile or using effective contraceptive with negative urinary pregnancy test

Part 2: Neuroendocrine tumor patients:

* Age between 18 and 75 years
* Signed Informed Consent
* Subject is diagnosed with a neuroendocrine tumor of gastroenteropancreatic, pulmonary, neural crest or unknown primary origin
* Subject is judged to be in good general condition by the investigator on the basis of medical history, physical examination including vital signs and clinical laboratory tests, besides the diagnosis of neuroendocrine tumor.
* Subject should have at least 5 positive lesions on routine clinical 68Ga-DOTA-peptide PET performed within 6 months prior to the inclusion visit. A positive lesion is defined as tracer uptake above background deemed to be caused by the presence of NET cells by an experienced nuclear medicine physician
* Female subjects should be post-menopausal or surgically sterile or using effective contraceptive with negative pregnancy test

Exclusion Criteria:

Part 1: Healthy volunteers:

* Subject has a previous or ongoing recurrent or chronic disease able to interfere with the evaluation of the trial according to the judgement of the investigator, especially a known gastro-intestinal, hepatic, renal, cardiovascular, metabolic or hormonal disease, cancer, major neurological or convulsive disorder or any psychiatric disease
* Subject is currently a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse
* Subject takes concomitant medication, except for oral contraceptives, sporadic paracetamol, or low-dose and limited in time non-steroidal antiinflammatory drugs
* Subject is unable to refrain from smoking more than 10 cigarettes per day during the study
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months
* Subject suffers from claustrophobia or cannot tolerate confinement during PET/CT scanning procedures; subject cannot lie still for 90 minutes inside the scanner
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e. weight lifting, running, bicycling) from the time of the selection visit until the safety visit
* Subject does not understand the study procedure
* Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator
* Subject is potentially pregnant (urinary hCG test will be performed in women where pregnancy is not excluded), wishes to become pregnant up to 3 months after administration of Al18F-NOTA-octreotide or is breast-feeding
* Subject has recently (< 30 days) participated or is simultaneously participating in another prospective interventional clinical trial
* Subject has a history of multiple and/or severe allergies to drugs or food
* Subject underwent surgery between the selection and inclusion visit
* Subject is mentally or legally incapacitated

Part 2: Neuroendocrine tumor patients:

* Subject has a previous or ongoing recurrent or chronic disease, other than a neuroendocrine tumor, at high risk to interfere with the evaluation of the trial according to the judgement of the investigator, e.g. known gastro-intestinal, hepatic, renal, cardiovascular, metabolic or hormonal disease, cancer, major neurological or convulsive disorder or any psychiatric disease
* Subject is currently a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse
* Subject is unable to refrain from smoking more than 10 cigarettes per day during the study
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months
* Subject suffers from claustrophobia or cannot tolerate confinement during PET/CT scanning procedures; subject cannot lie still for 60 minutes inside the scanner
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e. weight lifting, running, bicycling) from the time of the selection visit until the telephone follow-up interview.
* Subject does not understand the study procedure
* Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator
* Subject is potentially pregnant (urinary hCG test will be performed in women where pregnancy is not excluded), wishes to become pregnant up to 3 months after administration of Al18F-NOTA-octreotide or is breast-feeding
* Subject has recently (< 30 days) participated or is simultaneously participating in another prospective interventional clinical trial
* Subject has a history of multiple and/or severe allergies to drugs or food
* Subject underwent surgery between the selection and inclusion visit
* Subject is mentally or legally incapacitated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Potential of Al18F-NOTA-octreotide as somatostatin receptor PET imaging tracer in patients with neuroendocrine tumors | 1 year
  The primary endpoint will be met if in 4 out of 6 patients, at least two tumor lesions per patient are visualized in case of 5 to 10 known positive lesions on the 68Ga-DOTA-peptide PET, or at least 25% of the known tumor lesions per patient are visualized in case of more than 10 known positive tumor lesions on the 68Ga-DOTA-peptide PET. The study will be partially positive if in at least one patient at least 80% of the known positive lesions on the 68Ga-DOTA-peptide PET is visualized.

SECONDARY OUTCOMES:
Dosimetry of Al18F-NOTA-octreotide | 1 year
  Dosimetry will be assessed by means of the sequential whole-body PET/CT scans performed in healthy volunteers. Absorbed dose per unit of injected activity (mGy/MBq) at the organ and whole-body level will be calculated.
Normal-organ and tumor uptake of Al18F-NOTA-octreotide as a function of time | 1 year
  Patients will undergo dynamic PET scanning followed by three static whole-body PET/CT scans at different time points post injection. Uptake as a function of time (pharmacokinetics) will be studied using the software package PMOD (PMOD technologies LLC, Zürich, Switzerland). Volumes of interest (VOIs) will be delineated in relevant normal organs and tumor lesions on all PET images and standardized uptake values (SUV) in all these VOIs will be measured to compute normal-organ and tumor uptake as a function of time.
Identify the ideal time point for imaging after Al18F-NOTA-octreotide injection | 1 year
  Tumor-to-background ratios as a function of time will be measured. The time point resulting in optimal tumor-to-background ratios, taking into account a realistic implementation in clinical practice, will be defined as the ideal time point for imaging.
Safety analysis of Al18F-NOTA-octreotide administration: Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 1 year
  The impact of Al18F-NOTA-octreotide administration on clinical symptoms and signs and biochemistry values will be evaluated. Baseline values will be recorded and patients will be assessed clinically and with serial biochemical analysis. Adverse events will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Preliminary assessment of lesion targeting by Al18F-NOTA-octreotide as compared to 68Ga-DOTATATE | 1 year
  A lesion-by-lesion analysis (visual and semi-quantitative) will be performed to compare the number of detected lesions using both tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Deroose, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pauwels E, Cleeren F, Tshibangu T, Koole M, Serdons K, Dekervel J, Van Cutsem E, Verslype C, Van Laere K, Bormans G, Deroose CM. [18F]AlF-NOTA-octreotide PET imaging: biodistribution, dosimetry and first comparison with [68Ga]Ga-DOTATATE in neuroendocrine tumour patients. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3033-3046. doi: 10.1007/s00259-020-04918-4. Epub 2020 Jul 2. PMID 32617641